CLINICAL TRIAL: NCT01448915
Title: Management of Hepatitis C in HIV Infected IDUs
Brief Title: Management of Hepatitis C in HIV Infected Injection Drug Users (IDUs)
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: NA_00029706; R01DA016065 (NIH); NCT00496912 (obsolete NCT alias)
Record Dates: First submitted 2011-09-27; First posted 2011-10-07 (Estimated); Last update posted 2022-02-21 (Actual); Status verified 2021-02

CONDITIONS: HIV Infection; Hepatitis C
Keywords: HIV; Human immunodeficiency virus; Acquired Immune Deficiency Syndrome Virus; AIDS virus; Immunodeficiency Virus, Human; Virus, Human Immunodeficiency; Hepatitis C; Hepatitis C, chronic; Hepatitis C virus; Hepatitis C antibodies; Hepatitis C antigens
MeSH Terms: conditions — HIV Infections; Hepatitis C; Acquired Immunodeficiency Syndrome; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma specimens are collected at regular intervals
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons with HIV and HCV coinfection: Persons with HIV and HCV coinfection who receive medical care for HIV infection at Johns Hopkins Hospital

SUMMARY:
The principal goal of this research project is to evaluate the natural history of HCV and liver disease and its treatment in HIV-infected persons who use drugs. Research procedures will focus on determining liver disease prevalence and severity within this population. This is an observational study without study specific interventions.

DETAILED DESCRIPTION:
The principal goal of this research project is to evaluate the natural history of HCV and liver disease and its treatment in HIV-infected persons who use drugs. The recent availability of a novel, non-invasive method of measuring HCV disease stage makes it possible to test the relationship of HCV disease stage and the management of coinfected IDUs with adequate precision. The investigators will apply the innovative technology, elastography (FibroScan®) to ask whether the marked differences in the final disease outcome, end-stage liver disease (ESLD), can be explained by a measure of liver stiffness as assessed by elastography (FibroScan®). While advances in non-invasive disease assessment are critical to HCV management, the greatest challenge to improving HCV treatment effectiveness in coinfected persons remains low rates of treatment uptake and adherence, even when freely accessible. In response to this glaring disparity, the investigators will test potent behavioral reinforcement interventions to improve the management of HCV disease by adapting a rigorously studied contingent behavioral incentives program to the treatment to coinfected IDUs. Hepatitis C Treatment Eligibility: To determine the population prevalence of significant liver disease in coinfected IDUs using an innovative, non-invasive methodology (transient elastography, FibroScan®) to measure liver stiffness. Liver Disease Staging: To test the hypothesis that liver stiffness, assessed by a novel, non-invasive methodology, is predictive of the development of ESLD, defined as hepatic decompensation, hepatocellular cancer, and liver-related death, in coinfected IDUs.

ELIGIBILITY:
Inclusion Criteria:

* Current or prior drug use
* Reactive HCV antibody
* Reactive HIV antibody

Exclusion Criteria:

* Women may not undergo FibroScan while pregnant
* Persons with implanted cardiac devices may not undergo FibroScan

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational cohort of HIV-infected persons receiving medical care at the Johns Hopkins Hospital. Participants are eligible if they are HCV antibody positive and use or have used drugs.
Sampling Method: Non-Probability Sample
Enrollment: 828 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Hepatitis C Treatment Uptake and HCV cure | 5 years
  The proportion of persons with HIV and HCV coinfection who achieve HCV cure

SECONDARY OUTCOMES:
Incidence of clinical outcomes in persons with HIV/HCV coinfection with or without HCV cure | 5 years
  Clinical events including liver failure and liver cancer
Liver stiffness measurement by elastography in persons with HIV infection | 5 years
  Change in liver stiffness following HCV cure

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Sulkowski, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bilal U, Lau B, Lazo M, McCaul ME, Hutton HE, Sulkowski MS, Moore RD, Chander G. Interaction Between Alcohol Consumption Patterns, Antiretroviral Therapy Type, and Liver Fibrosis in Persons Living with HIV. AIDS Patient Care STDS. 2016 May;30(5):200-7. doi: 10.1089/apc.2016.0010. PMID 27158847
- [Result] Falade-Nwulia O, Sutcliffe C, Moon J, Chander G, Wansom T, Keruly J, Katzianer J, Nathanson A, Marks J, Mehta S, Thomas D, Moore R, Sulkowski M. High hepatitis C cure rates among black and nonblack human immunodeficiency virus-infected adults in an urban center. Hepatology. 2017 Nov;66(5):1402-1412. doi: 10.1002/hep.29308. Epub 2017 Oct 11. PMID 28608973
- [Result] Wansom T, Falade-Nwulia O, Sutcliffe CG, Mehta SH, Moore RD, Thomas DL, Sulkowski MS. Barriers to Hepatitis C Virus (HCV) Treatment Initiation in Patients With Human Immunodeficiency Virus/HCV Coinfection: Lessons From the Interferon Era. Open Forum Infect Dis. 2017 Feb 11;4(1):ofx024. doi: 10.1093/ofid/ofx024. eCollection 2017 Winter. PMID 28480293